CLINICAL TRIAL: NCT06827938
Title: Multicenter Real-World Study of Hyperthermia in Skin/Mucosal HPV Infection of Special Population
Brief Title: Multicenter Real-World Study of Hyperthermia in Warts of Special Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, Professor, First Hospital of China Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF-SOP-07-1.2-01
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Warts
Keywords: warts; local hyperthermia
MeSH Terms: conditions — Warts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperthermia group (Other): Infrared hyperthermia（44±1℃） device for 3 consecutive days (times / day), each treatment for 30 minutes After 7-10 days, the lesions of the same target were treated continuously for 2 days (times / day), and then treat every 7-10 days, the method was the same as before. Lesion changes were assessed after 15 treatments.
  Interventions: Device: YY-WRY-V01 Infrared thermotherapy apparatus

INTERVENTIONS:
Device: YY-WRY-V01 Infrared thermotherapy apparatus — Infrared hyperthermia（44±1℃） device for 3 consecutive days (times / day), each treatment for 30 minutes After 7-10 days, the lesions of the same target were treated continuously for 2 days (times / day), and then treat every 7-10 days, the method was the same as before. Lesion changes were assessed after 15 treatments.

SUMMARY:
Hyperthermia refers to treating diseases with temperatures beyond normal body temperature (39-45℃), and moxibustion therapy of traditional Chinese medicine belongs to the category of hyperthermia. It has been reported at home and abroad that the local temperature of 44℃ can effectively mobilize the body's immunity and remove HPV infection lesions, such as condyloma acuminatum and verruca vulgaris. Our research group conducted randomized controlled experiments on patients with viral warts in the early clinical practice, and the cure rate of the hyperthermia group reached 45-55%, which was superior to the traditional method in the aspects of no trauma, low recurrence rate, easy to tolerate and so on. Our research group's preliminary research on hyperthermia of viral warts has been included in the British Medical Association's guidelines for viral warts therapy. The equipment our research group developed has been obtained the medical device registration certificate, and is in the process of national promotion. Hyperthermia is to mobilize systemic immunity through local warm heat, the preliminary clinical study of the research group shows that the therapeutic effect of hyperthermia is usually "all or none": "all" that is, after hyperthermia, all viral warts are removed, including non-treatment lesions;"None" means that some patients with viral warts do not respond to hyperthermia. Cellular immunity plays a very important role in the removal of warts. At present, some special clinical patients such as pregnant women, children, patients with autoimmune diseases, diabetes, immunosuppressants after organ transplantation and other patients with skin/mucosal HPV infection, their warts show more extensive proliferation or a longer and repeated course of disease, treatment resistance, etc. It has increased the difficulty of clinical treatment, and the specific mechanism is still unclear. Therefore, for these special populations, how to further enhance the therapeutic effect of hyperthermia is the top priority of current research.

In view of the above findings, this research group intends to study the efficacy and safety of hyperthermia in the treatment of viral warts in the special population (pregnant women, children, patients with autoimmune diseases, diabetes, and immunosuppressants after organ transplantation, etc.) in a multicenter real-world study of skin/mucosal HPV infection in the special population.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with viral warts
2. Diagnosis of AIDS with viral warts
3. Autoimmune disease patients with viral warts
4. Diabetic patients with viral warts
5. Patients with viral warts who are currently being treated with immunosuppressants
6. Children with viral warts
7. The subject or legal guardian is able to understand and sign the informed consent/consent to participate in the study

Exclusion Criteria:

1. The subject suffers from tumor or other serious disease and cannot complete this clinical study
2. Timely treatment and follow-up cannot be guaranteed due to personal or other objective reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
The cure rate | Three months
  Three months after treatment, the overall cure rate of skin lesions is assessed.
The cure rate | Six months
  Six months after treatment, the overall cure rate of skin lesions is assessed.
The recurrence rate | Three months
  Three months after treatment, the recurrence rate of skin lesions is assessed.
The recurrence rate | Six months
  Six months after treatment, the recurrence rate of skin lesions ie assessed.

SECONDARY OUTCOMES:
The rate of adverse reaction | Three months
  During treatment, adverse reactions and the incidence of treatment-related adverse reactions were recorded.
The rate of adverse reaction | Six months
  During treatment, adverse reactions and the incidence of treatment-related adverse reactions were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No